CLINICAL TRIAL: NCT05565118
Title: Prospective Surgical Study on the Pattern of Electrical Activity in High Grade Glioma (WHO Grade III and IV) as a Predictor of Progression
Brief Title: Prospective Surgical Study on the Pattern of Electrical Activity in High Grade Glioma as a Predictor of Progression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Burkhardt Brain Tumor and Neuro-Oncology Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4321
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: High Grade Glioma; Glioblastoma
Keywords: High Grade Glioma; Glioblastoma; Neural Recording; Electrical Activity
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Intervention Model Description: Participants undergoing surgical resection will have a regional recording of neuronal electrical activity that will be measured in a minimum of 4 peritumoral anatomic zones via depth electrodes, overlying the cortex of the lesion via a subdural grid, within the presumed tumor, and in adjacent presumed normal brain. Recording findings specific to these anatomo-electro-clinical zones will be correlated with the presence/degree of contrast-enhancing tumor on MRI at recurrence. Additionally, biopsies will be obtained in these depth electrode regions for correlative studies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard Surgical Treatment + Intraoperative Electrocorticography (Experimental): Each participant will undergo intraoperative electrocorticography (ECOG) through subdural grid (SDG) and depth electrode (DE) via FDA-cleared, standardized, brain recording technology. During this surgery, participants will also undergo a tissue biopsy at recording sites for correlation to neural recording data.
  Interventions: Procedure: Standard Surgical Treatment; Procedure: Intraoperative Electrocorticography

INTERVENTIONS:
Procedure: Standard Surgical Treatment — During this surgery, participants will also undergo a tissue biopsy at recording sites for correlation to neural recording data.
Procedure: Intraoperative Electrocorticography — Each participant will undergo intraoperative electrocorticography (ECOG) through subdural grid (SDG) and depth electrode (DE) via FDA-cleared, standardized, brain recording technology.

SUMMARY:
The purpose of this study is to test the safety and feasibility of recording brain activity within and around high-grade glioma tumors at the time of surgery. A small biopsy will be taken at the sites of the recordings.

DETAILED DESCRIPTION:
High-grade gliomas are incurable primary brain tumors. Recent data support that glioma cells can integrate within neuronal circuits. Glioma cells and neurons communicate via electrical impulses and chemically, through neurotransmitters. This crosstalk has been shown to promote glioma cell migration and invasion in preclinical models. However, the nature of the electrical activity and underlying molecular mechanisms are poorly understood. The long-term goal of this study is to determine the impact of high electrical activity and pattern of activity on tumor invasion, and mechanistic basis of its regulation and functional consequences. This phase I safety and feasibility study is being proposed as a first step toward dissecting the connection between electrical activity and glioma behavior. The goal is to determine the safety and feasibility of recording electrical activity in the tumor-neuron interface using technologies that are already being used clinically for participants undergoing brain surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have the appearance of high-grade glioma (HGG, WHO Grade 3 and 4, including GBM) on MR imaging are allowed to consent and will undergo the procedure if the frozen is consistent with HGG

OR

* Participants with a history of histologically-confirmed diagnosis of high- grade glioma that are undergoing resection of a recurrent/progressive tumor that is likely recurrent/progressive high- grade glioma as identified on preoperative MR imaging
* Age ≥ 18 years old
* Volumetric MRI within 1 month prior to surgery
* Karnofsky performance status of 60 or higher
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Participants must be considered appropriate neurosurgical candidates with the following screening/baseline laboratory values within 1 month prior to surgery:

  * Absolute neutrophil count ≥ 1500/µL
  * Platelets ≥ 100 000/µL
  * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × Upper limit of normal (ULN) unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
  * Urine or Serum Pregnancy Test = Negative (Not applicable to participants with bilateral oophorectomy and/or hysterectomy or to those participants who are postmenopausal).

Exclusion Criteria:

* Severe co-morbidity that would confer excess risk of surgery as determined by the treating physician.
* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
* Is pregnant
* Coagulopathy or platelet dysfunction that increases the risk of intra and postoperative hemorrhage
* Tumor location requiring DE placement/biopsy in eloquent or critical region of the brain (e.g. primary motor and sensory cortices, speech and vision centers, thalamus, basal ganglia, cerebellum, brain stem) as deemed by the neurosurgeon designing the surgical plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between electrical activity and anatomic region of progression based on follow-up contrast-enhanced MRI | Up to 9 months post surgery
  To describe the pattern of electrical activity (neuronal hyperexcitability) in brain surrounding the enhancing tumor during open surgery in patients with high grade gliomas and its correlation with progression

OTHER OUTCOMES:
Correlation between electrical activity (neuronal hyperexcitability) in brain surrounding the enhancing tumor and cellular and molecular profile of the tumor and its microenvironment | At study completion, an aim for 1 year post treatment
  Electrical activity will be assessed as described above and correlated with transcriptomic changes. Bioinformatics analyses including gene ontology analyses and multi-dimensional network analyses will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Yu, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared, while individual data will not need to be shared.